CLINICAL TRIAL: NCT06164171
Title: Transesophageal Echocardiography (TEE) and Simulation : a Preferred Learning Path
Acronym: TEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7646
Record Dates: First submitted 2022-11-08; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Disease
Keywords: Cardiac disease; Transesophageal echocardiography; TEE; High definition simulator
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transesophageal echocardiography (TEE) has gradually become the technique of choice for continuous functional examination of the heart despite the significant training required for its interpretation. It has proven to be the safest, fastest, and most reliable technique for diagnosing most intra- and postoperative hemodynamic problems. Indeed, the transesophageal route is particularly well adapted to the situation of intubated patients, whether in the operating room, in the outpatient department or in intensive care. It offers images that are easier to obtain and of better quality than the transthoracic route; it can be performed without interfering with surgical activity or resuscitation. However, TEE training is often poor during the DES training in anesthesia and resuscitation, reserved for the few interns who will learn in a specific department where TEE is used on a daily basis.

Thus, simulation is a logical and recognized means by which technical aspects, mechanisms involved in the understanding of a situation, reasoning and decision making can be analyzed and improved.

The RFE SFAR 2019 recommendations suggest the use of simulation for the learning of technical gestures in initial training in order to improve their acquisition.

This study is therefore part of a technical and diagnostic improvement of a practice, which appears to be essential in several fields in anesthesia and intensive care, for a technique still not sufficiently acquired by many future practitioners.

ELIGIBILITY:
Inclusion criteria:

* 1st or 2nd year DESAR interns who participated in the continuing education program
* Interns who agreed to participate in the professional practice evaluation study

Exclusion criteria :

* Interns who did not participate in the training
* Residents who do not agree to take the final test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1st or 2nd year DESAR interns who participated in the continuing education program
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability of a population of medical students to perform a TEE thanks to the contribution of simulation to their learning compared to a population of interns not trained on a high definition simulator Time in seconds required to make the 11 cuts | 1 hour after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France